CLINICAL TRIAL: NCT07002632
Title: Effect of Preoperative Dexpanthenol Moisturizer on the Prevention of Angular Cheilitis After Pediatric Adenotonsillectomy: A Randomized Controlled Trial
Brief Title: Using Dexpanthenol Cream to Prevent Lip Corner Cracks in Children After Tonsil/Adenoid Surgery
Acronym: PrevAC-PedAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 309 Anguler Cehilitis
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cheilitis, Angular; Postoperative Complications; Adenotonsillar Hypertrophy
Keywords: Cheilitis, Angular; Tonsillectomy; Adenoidectomy; Dexpanthenol; Pain; Pediatrics
MeSH Terms: conditions — Cheilitis; Postoperative Complications; Pain | interventions — dexpanthenol; Ointments

STUDY DESIGN:
Intervention Model Description: This was a parallel-group, randomized, controlled trial. Participants were randomly assigned to one of two arms: an intervention group receiving preoperative dexpanthenol moisturizer or a control group receiving no preoperative topical intervention. Participants remained in their assigned group for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor, a senior surgeon responsible for evaluating postoperative angular cheilitis and pain, was blinded to the treatment group allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexpanthenol group (Experimental): Participants in this arm received a single application of 5% dexpanthenol cream (water-in-oil emulsion) to both oral commissures. The cream was applied immediately before mouth gag insertion at the start of the adenotonsillectomy procedure.
  Interventions: Drug: Dexpanthenol 5 % Topical Ointment
- Control group (No Intervention): Participants in this arm received no topical cream or moisturizer on the oral commissures before or during the adenotonsillectomy procedure.

INTERVENTIONS:
Drug: Dexpanthenol 5 % Topical Ointment — Dexpanthenol is a topical agent, a derivative of pantothenic acid (a B-complex vitamin), used for its moisturizing and skin regenerative properties. The formulation studied was a 5% dexpanthenol in a water-in-oil emulsion.
  Other Names: Bepanthol Derma moisturizing cream
  Arms: Dexpanthenol group

SUMMARY:
Soreness and cracking at the corners of the mouth, a condition called angular cheilitis, can be an uncomfortable problem for children after they have surgery to remove their tonsils and adenoids. This study looks at whether applying a moisturizing cream containing dexpanthenol to the corners of the mouth right before the surgery can help prevent this from happening.

The main idea (hypothesis)i the investigators are testing is that this dexpanthenol cream will protect the skin and reduce the number of children who get these painful lip sores after their operation.

To find this out, children who are scheduled to have tonsil and/or adenoid surgery will be invited to join the study. Children (participants) will be randomly placed into one of two groups by chance. One group of children will have the dexpanthenol cream applied to their lip corners just before their surgery. The other group will not have any cream applied to their lip corners before surgery. After the surgery, investigators will check all children to see if they have developed lip corner sores and compare how many children in each group experienced this problem.

The goal of this research is to see if this simple cream application can be an easy way to help children feel more comfortable while they are recovering from their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 15 years, inclusive
* Scheduled for adenotonsillectomy (for indications such as obstructive sleep apnea and/or recurrent tonsillitis/adenotonsillitis).
* Written informed consent provided by parents or legal guardians.

Exclusion Criteria:

* Known allergy or hypersensitivity to dexpanthenol or any components of the cream.
* Presence of angular cheilitis at the time of preoperative assessment.
* Use of topical or systemic steroids or antibiotics within 4 weeks prior to surgery that might affect oral healing.
* Participants with known systemic diseases or conditions that might impair wound healing (e.g., uncontrolled diabetes, immunosuppressive disorders).
* Known diagnosis of iron deficiency and/or vitamin B12 deficiency prior to surgery.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ethem ilhan, MD, Principal Investigator — Department of ENT, University of Health Sciences, Gaziosmanpasa TREH, Istanbul, Turkey
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] England RJ, Lau M, Ell SR. Angular cheilitis after tonsillectomy. Clin Otolaryngol Allied Sci. 1999 Aug;24(4):277-9. doi: 10.1046/j.1365-2273.1999.00255.x. PMID 10472460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Department of Otorhinolaryngology at a single tertiary care center, Gaziosmanpasa Training and Research Hospital, in Istanbul, Turkey. The recruitment period for the study was between July 2021 and June 2024. Eligible participants were children aged 3 to 15 years who were scheduled for adenotonsillectomy and were identified during their routine preoperative clinical assessment.
Pre-assignment Details: No pre-assignment events, such as a run-in or washout period, occurred in this study. Enrolled participants were directly randomized to their assigned group after meeting the eligibility criteria.
Period: Overall Study
Arm/Group | Dexpanthenol Group | Control Group
Started | 53 | 53
Completed | 51 | 50
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: A total of 106 participants were initially enrolled and randomized into the study. However, five participants were lost to follow-up and their data were excluded from the final analysis. Therefore, the baseline characteristics are reported for the 101 participants who completed the study and were included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexpanthenol Group | Control Group | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.65 (2.36) | 5.96 (2.82) | 6.31 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 26 | 30 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 51 | 50 | 101
Pre-operative Tonsil Grade [Count of Participants; unit: Participants] — Pre-operative tonsil grade was assessed using the Brodsky grading scale. This clinical scale categorizes tonsil size based on the proportion of the oropharyngeal airway occupied by the tonsils: Grade 1 = <25%, Grade 2 = 25-50%, Grade 3 = 50-75%, and Grade 4 = >75%. Higher grades indicate more severe tonsillar hypertrophy.
  Participants
    Grade 1 | 8 | 7 | 15
    Grade 2 | 14 | 14 | 28
    Grade 3 | 18 | 16 | 34
    Grade 4 | 11 | 13 | 24
Surgical Indication [Count of Participants; unit: Participants]
  Obstructive sleep apnea | 14 | 13 | 27
  Recurrent adenotonsillitis | 10 | 6 | 16
  Recurrent tonsillitis + obstructive sleep apnea | 27 | 31 | 58
Mallampati Classification [Count of Participants; unit: Participants] — Mallampati classification was used to assess the visibility of oropharyngeal structures when the patient opened their mouth and protruded the tongue. The scale includes four classes:
  * Class I: soft palate, uvula, fauces, and tonsillar pillars are visible;
  * Class II: soft palate, uvula, and fauces are visible;
  * Class III: only soft palate and base of the uvula are visible;
  * Class IV: only the hard palate is visible. Lower classes indicate a wider oropharyngeal space, while higher classes represent more restricted visibility."
  Participants
    class 1 | 43 | 39 | 82
    class 2 | 8 | 11 | 19
    class 3 | 0 | 0 | 0
    class 4 | 0 | 0 | 0
Vertical mouth opening length [Mean (Standard Deviation); unit: centimeters] | 4.48 (0.70) | 4.63 (0.89) | 4.55 (0.80)
Mouth opener size [Mean (Standard Deviation); unit: centimeters] | 7.36 (0.76) | 7.01 (1.15) | 7.18 (0.98)
Operation time [Mean (Standard Deviation); unit: minutes] | 35.10 (14.39) | 38.86 (18.53) | 36.96 (16.59)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Angular Cheilitis
Description: Presence or absence of angular cheilitis determined by clinical examination. Angular cheilitis was defined as any inflammation, erythema, fissures, ulceration, or crusting at one or both oral commissures. Evaluations were performed by a senior surgeon blinded to treatment group allocation.
Time Frame: Postoperative Day 1 and Postoperative Day 7
Population: The analysis for this outcome measure was performed on all participants who completed the study. A total of 106 participants were initially randomized, but five were lost to follow-up. Therefore, the analysis population for this outcome consists of the 101 participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpanthenol Group | Control Group
Number analyzed (Participants) | 51 | 50
Participants
  1st day Angular cheilitis pozitif | 5 | 22
  1st day Angular cheilitis negative | 46 | 28
  1st week Angular cheilitis pozitif | 2 | 5
  1st week Angular cheilitis negative | 49 | 45

2. Secondary Outcome: Postoperative Pain Score
Description: Pain intensity was assessed by the parents using the Wong-Baker FACES Pain Rating Scale. The scale ranges from 0 (no hurt) to 10 (hurts worst).
Time Frame: Postoperative Day 1 and Postoperative Day 7
Population: The analysis for this outcome measure was performed on all participants who completed the study. A total of 106 participants were initially enrolled, but five were lost to follow-up. Therefore, the analysis population for this outcome consists of the 101 participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexpanthenol Group | Control Group
Number analyzed (Participants) | 51 | 50
score on a scale
  1st day pain score | 4.47 (1.93) | 4.48 (1.94)
  1st week pain score | 2.41 (1.66) | 2.38 (1.59)

ADVERSE EVENTS:
Time Frame: From the day of surgery to the final study follow-up on the seventh postoperative day.
Description: The systematic assessment was limited to the pre-specified primary outcome (incidence of angular cheilitis) and secondary outcome (postoperative pain). No other adverse events were systematically monitored or recorded as part of the study protocol.
Arm/Group | Dexpanthenol Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 51/51 | 50/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexpanthenol Group (N=51) | Control Group (N=50)
Angular Cheilitis (Skin and subcutaneous tissue disorders) | 5 (5) | 22 (22) — Localized inflammation, erythema or crusting at the corner of the mouth
Postoperative Pain (General disorders) | 51 (51) | 50 (50) — Pain was evaluated using the Wong-Baker FACES Pain Rating Scale (0-10) on postoperative days 1 and 7. All participants reported some level of postoperative pain, which was expected and non-serious.

LIMITATIONS AND CAVEATS:
A precise a priori power analysis was not feasible due to limited prior literature. The study's single-center design may limit the generalizability of the findings. The short, seven-day follow-up period does not allow for assessment of long-term effects. Finally, the parent-reported rating scale for the secondary outcome of pain introduces a degree of subjectivity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT07002632/Prot_SAP_000.pdf